CLINICAL TRIAL: NCT03671967
Title: Piperacillin Tazobactam Versus Meropenem for Treatment of Bloodstream Infections Caused by Cephalosporin-resistant Enterobacteriaceae- a Non-inferiority Randomized Controlled Trial
Brief Title: PipEracillin Tazobactam Versus mERoPENem for Treatment of Bloodstream Infections Caused by Cephalosporin-resistant Enterobacteriaceae (PETERPEN)
Acronym: PETERPEN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Rabin Medical Center (Other); University of Modena and Reggio Emilia (Other); Tel Aviv Medical Center (Other); Meir Medical Center (Other); Soroka University Medical Center (Other); The Chaim Sheba Medical Center (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Jewish General Hospital (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOH_2018-12-25_004857
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Beta Lactam Resistant Bacterial Infection; Enterobacteriaceae Infections; Bacteremia
Keywords: bacteremia; enterobacteriaceae; extended spectrum beta-lactamase; meropenem; piperacillin tazobactam
MeSH Terms: conditions — Enterobacteriaceae Infections; Bacteremia | interventions — Piperacillin, Tazobactam Drug Combination; Meropenem

STUDY DESIGN:
Intervention Model Description: open-label randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- piperacillin tazobactam (Experimental)
  Interventions: Drug: Piperacillin/tazobactam
- meropenem (Active Comparator)
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Piperacillin/tazobactam — 4.5 grams QID
  Arms: piperacillin tazobactam
Drug: Meropenem — 1 gram TID
  Arms: meropenem

SUMMARY:
Data regarding optimal treatment for extended-spectrum beta-lactamase (ESBL) producing Enterobacteriaceae blood-stream infection are lacking. Observational studies show conflicting results when comparing treatment with combination beta-lactam-beta-lactamase inhibitor and carbapenems. The investigators aim to evaluate the effect of definitive treatment with meropenem vs. piperacillin-tazobactam on the outcome of patients with bacteremia due to cephalosporin-non-susceptible Enterobacteriaceae. The investigators hypothesize that piperacillin-tazobactam is non-inferior to meropenem.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age ≥ 18 years)
2. New onset BSI due to E. coli or Klebsiella spp. in one or more blood cultures associated with evidence of infection.
3. The microorganism will have to be non-susceptible to third generation cephalosporins (ceftriaxone and ceftazidime) and susceptible to both PTZ and meropenem (see microbiological methods).
4. Both community and hospital-acquired bacteremias will be included.
5. We will permit the inclusion of bacteremias due to E. coli or Klebsiella spp. with concomitant growth in blood of skin commensals considered as contaminants.

Exclusion Criteria:

1. More than 72 hr. elapsed since initial blood culture taken, regardless of the time covering antibiotics were started (up to 72 hrs.).
2. Polymicrobial bacteremia. Polymicrobial bacteremia will be defined as either growth of two or more different species of microorganisms in the same blood culture, or growth of different species in two or more separate blood cultures within the same episode.
3. Patients with prior bacteremia or infection that have not completed antimicrobial therapy for the previous infectious episode.
4. Patients with septic shock at the time of enrollment and randomization, defined as at least 2 measurements of systolic blood pressure < 90 mmHg and/or use of vasopressors (dopamine>15μg/kg/min, adrenalin>0.1μg/kg/min, noradrenalin>0.1μg/kg/min, vasopressin any dose) in the 12 hours prior to randomization. In the absence of the use of vasopressors, a systolic blood pressure <90 would need to represent a deviation for the patient's known normal blood pressure.
5. BSI due to specific infections known at the time of randomization:

   1. Endocarditis / endovascular infections
   2. Osteomyelitis (not resected)
   3. Central nervous system infections
6. Allergy to any of the study drugs confirmed by history taken by the investigator
7. Previous enrollment in this trial
8. Concurrent participation in another interventional clinical trial
9. Imminent death (researcher's assessment of expected death within 48 hrs. of recruitment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1084 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 30 days from randomization
Treatment failure | 7 days from randomization
  death OR fever > 38°C in the last 48 hours OR lack of resolution of symptoms attributed to the focus of infection OR Sequential Failure Organ Assessment (SOFA) score increasing OR positive blood cultures by the time point assessed

SECONDARY OUTCOMES:
All-cause mortality | 14 and 90 days from randomization
Treatment failure | 14 days and 30 days from randomization
  death OR fever > 38°C in the last 48 hours OR lack of resolution of symptoms attributed to the focus of infection OR Sequential Failure Organ Assessment (SOFA) score increasing OR positive blood cultures by the time point assessed
Microbiological failure | 7 days and 14 days from randomization
  Repeat positive blood cultures with index pathogen on day 4 or later from randomization
Recurrent positive blood cultures (relapse) | 30 days and 90 days from randomization
  recurrent positive blood cultures with the index pathogen after prior sterilization of blood cultures or after end of treatment
Clostridium difficile associated diarrhea | 90 days from randomization
Clinically or microbiologically documented infection other than Gram-negative bacteremia | 90 days from randomization
Number of hospital re-admissions | 90 days from randomization
Development of resistance | 90 days from randomization
  clinical isolates resistant to piperacillin/tazobactam and meropenem and any carbapenem-resistant bacteria
Carriage of carbapenemase-producing Enterobacteriaceae (CPE) and non-CPE carbapenem-resistant Enterobacteriaceae in-hospital | 90 days from randomization
  detected by weekly rectal surveillance of carriage while in-hospital
Total in-hospital days | 30 days and 90 days from randomization
Total antibiotic days | 30 days and 90 days from randomization
Adverse events | 30 days from randomization
  diarrhea, liver function test abnormalities, antibiotic rash or other immediate-type allergy, acute kidney injury defined according to RIFLE criteria

CONTACTS AND LOCATIONS:
Overall Officials: Roni Bitterman, MD, Principal Investigator — Rambam Health Care Campus; Mical Paul, MD, Study Director — Rambam Health Care Campus; Leonard Leibovici, MD, Study Director — Rabin Medical Center; Cristina Mussini, MD, Study Director — University of Modena and Reggio Emilia; Noa Eliakim-Raz, MD, Study Director — Rabin Medical Center, Beilinson Campus
Locations (14):
- Canada (6):
  - University of Calgary, Cumming School of Medicine, O'Brien Institute for Public Health, Calgary, Alberta
  - Surrey Memorial Hospital - Fraser Health Authority, Surrey, British Columbia
  - Eastern Health, St. John's, Newfoundland and Labrador
  - Kingston General Hospital, Kingston, Ontario
  - Jewish Genral Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
- Israel (8):
  - Rambam Health Care Campus, Haifa, Israel
  - Soroka Medical Center, Beersheba
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Sanz Medical Center-Laniado Hospital, Netanya
  - Rabin Medical Center, Beilinson Campus, Petah Tikva
  - Sheba Medical Center (Tel HaShomer), Tel Aviv
  - Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data collected during the trial will be made available for an unlimited time period following publication of trial results. Data will be available for researchers who provide a methodologically sound proposal and contingent on both the researchers' and our ethics committee approval and the signing of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: following publication and for unlimited time
Access Criteria: proposals should be sent to the principal investigator at ro_oren@rambam.health.gov.il

REFERENCES:
- [Derived] Bitterman R, Koppel F, Mussini C, Geffen Y, Chowers M, Rahav G, Nesher L, Ben-Ami R, Turjeman A, Huberman Samuel M, Cheng MP, Lee TC, Leibovici L, Yahav D, Paul M. Piperacillin-tazobactam versus meropenem for treatment of bloodstream infections caused by third-generation cephalosporin-resistant Enterobacteriaceae: a study protocol for a non-inferiority open-label randomised controlled trial (PeterPen). BMJ Open. 2021 Feb 8;11(2):e040210. doi: 10.1136/bmjopen-2020-040210. PMID 33558347